CLINICAL TRIAL: NCT04047849
Title: The Effect of Antibiotics on Latency in Previable Prelabor Rupture of Membranes Between 18 0/7 and 22 6/7 Weeks Gestational Age
Brief Title: Latency Antibiotics in Previable PPROM, 18 0/7- 22 6/7 WGA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-19-001
Record Dates: First submitted 2019-07-10; First posted 2019-08-07 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Rupture of Membranes; Delayed Delivery (Following Spontaneous Rupture); Rupture of Membranes; Premature; Rupture of Membranes; Premature, Affecting Fetus; Preterm Birth; Preterm PROM (Pregnancy); Preterm Labor
Keywords: Previable; PPROM; Premature prelabor rupture of membranes; Preterm; Preterm birth; Latency antibiotics
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Premature Birth; Obstetric Labor, Premature; Preterm Premature Rupture of the Membranes | interventions — Anti-Bacterial Agents; Azithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: The treatment group will include those subjects randomized to the antibiotic arm versus the control arm, no antibiotics. The antibiotic arm will receive a single, 500mg dose of Azithromycin given prior to discharge to home, followed by 250mg daily for 4 more days, and Amoxicillin 500mg orally TID for 7 days (first dose also being given prior to discharge home). Both arms will receive patient pamphlets with study contacts, precautions, and graphs for daily temperature/symptom tracking. Weekly follow up with Maternal-Fetal Medicine, for both arms, will include history and physical exam, vital signs, and ultrasound for fetal well-being and measurement of AFI. Both arms will be re-admitted to the hospital either at 1) viability (23 0/7 weeks) or 2) clinical signs of placental abruption, preterm labor, chorioamnionitis or fetal demise. Re-admission of both arms at viability will include latency antibiotics, neuroprotective magnesium sulfate, and corticosteroids for fetal lung maturity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antibiotics (Experimental): This will include those subjects randomized into the treatment arm, receiving the outpatient antibiotic course of azithromycin and amoxicillin prior to re-admission at viability (23 0/7 weeks gestation). They will receive a single, 500mg dose of Azithromycin given prior to discharge to home, followed by 250mg daily for 4 more days, and Amoxicillin 500mg orally TID for 7 days (first dose also being given prior to discharge home).
  Interventions: Drug: Antibiotics, oral Azithromycin and oral Amoxicillin
- No antibiotics (No Intervention): This will include those subjects randomized into the control arm and will not receive outpatient antibiotics prior to re-admission at viability (23 0/7 weeks gestation).

INTERVENTIONS:
Drug: Antibiotics, oral Azithromycin and oral Amoxicillin — Azithromycin (500mg day one followed by 250mg per day for 4 more days) and amoxicillin (500mg orally three times daily for 7 days) for a total course of seven days of antibiotic therapy
  Other Names: Z-pack
  Arms: Antibiotics

SUMMARY:
This study is a non-blinded, prospective, randomized controlled trial designed to compare the effect of outpatient oral antibiotics (i.e., amoxicillin and azithromycin) on the length of time (days) that pregnancy continues after a patient's water bag has ruptured prematurely. If a patient has been diagnosed with rupture of their water bag between 18 0/7 weeks and 22 6/7 weeks and there are no other associated complications with the pregnancy, the patient is eligible for initial consideration for this study. Patients will be admitted to the hospital for a 24-hour monitoring period. If the patient remains without further complications during this monitoring period, the patient will be eligible for enrollment. If enrollment is desired, the patient will be randomly assigned to receive either antibiotics (treatment arm of the study) or no antibiotics (control arm of the study). The treatment arm will receive an outpatient, 7-day course of oral antibiotics (azithromycin and amoxicillin) with the first dose given in the hospital to ensure no side effects. The control arm will not receive outpatient antibiotics. Both groups will have weekly, office follow-up visits with high-risk pregnancy specialists to ensure no further complications. Both groups will be admitted to the hospital if the patients reach 23 0/7 weeks without complications. At this time the patients will receive all medications and therapies recommended by the governing board of OBGYNs. Subjects of both groups will also be admitted before 23 0/7 weeks if further complications noted either at their clinic follow up visits or anytime outside of the hospital. The duration of time that the patient remains pregnant after breaking of the water bag will be compared in each group. The investigators will also see if there is a difference in the number of patients able to reach 23 0/7 weeks between each group (treatment versus control).

DETAILED DESCRIPTION:
Throughout this detailed description, patient and subject will be used interchangeably.

Patients presenting to either an acute care setting (Woman's Hospital Assessment Center) or outpatient clinic setting with concerns for rupture of membranes will be clinically evaluated by an obstetrician (including private physicians, resident faculty and resident physicians). Exam findings including either/or 1) visualization of amniotic fluid passing from the cervical canal and pooling in the vagina via sterile speculum examination, 2) a basic pH (i.e., positive nitrazine) test of vaginal fluid, 3) arborization (ferning) of dried vaginal fluid identified via microscopic examination by the examining physician, or 4) an amniotic fluid index (AFI) of less than 4cm between 18 0/7 and 22 6/7 weeks gestation are to be diagnostic of previable, preterm premature rupture of membranes (PPROM). Eighteen weeks gestational was arbitrarily chosen as the lower limit of gestational ages included based on review of currently available retrospective studies on previable PPROM. If patient meets all inclusion and exclusion criteria as listed above specimens to be collected at the time of diagnosis include a catheterized urinalysis with reflex urine culture if indicated, wet prep (i.e., vaginitis panel), group B strep DNA recto-vaginal swab, complete blood count and PCR testing for gonorrhea, chlamydia and trichomonas via endocervical swab. An ultrasound to determine amniotic fluid index (AFI) should also be performed at this time (either by radiology or Maternal-Fetal Medicine). These will be collected according to current standard of care practices for preterm prelabor rupture of membranes. Patient will then be admitted to the Woman's Hospital Labor and Delivery unit for a 24-hour observation period. Acetaminophen and ibuprofen will be withheld during this 24-hour observation period in order to ensure that no signs or symptoms of underlying infection or preterm labor are masked. A repeat complete blood count will be performed the morning of hospital day 2, and repeat AFI on hospital day 2 to be performed with full obstetric ultrasound by Maternal Fetal medicine physicians.

If, during the 24-hour observation period, the subject is without signs of chorioamnionitis, preterm labor, or placental abruption with vaginal bleeding as determined by the MFM staff, and if patient continues to meet both inclusion and exclusion criteria, subject will then be offered enrollment in the study. The consenting process will be performed by the MFM staff physicians or by Felicia LeMoine, MD, or Kaitlyn Taylor, MD, the co-investigators. The consenting process will be performed within the patient's private hospital room (designated at the time of admission). Once the subject as agreed to voluntary participation and in-formed consent has been signed, the subject will then be assigned an individual study identifier that includes the study acronym OAPPPROM patient initials, and unique number (randomly generated using the sample () function in R statistical software). All blood samples and specimens collected prior to admission, at admission and future blood samples and specimens will be available to the treating physician and reported within the patient's chart as is current standard practice. The samples and specimens will also be referenced using the patient's unique identifier for the sake of research data collection. The enrolled subjects will then be randomized using a computer-generated sample without replacement from the patient ID numbers into either the control (no antibiotics) or treatment (antibiotics) arm.

Following the 24-hour observation period and randomization, those subjects enrolled into the treatment (antibiotics) arm of the study will be thoroughly counseled on the risks and adverse side effects associated with the use of azithromycin and amoxicillin and which of those side effects should prompt emergency evaluation at Woman's Hospital Assessment Center or the nearest emergency department with obstetrical care. The subjects of the treatment arm will also receive the first dose of antibiotics while in the hospital to ensure no immediate adverse effects.

Both arms of the study will receive, at the time of discharge, a "Patient Information Pamphlet" along with a thermometer to take home. All subjects will be instructed on proper methods to measure body temperature with the thermometer. All subjects will be thoroughly counseled on symptoms or findings which should prompt immediately follow-up at Woman's Hospital or the nearest emergency department with obstetrical care. Such symptoms include, but are not limited to, vaginal bleeding, fevers, chills, purulent vaginal discharge, contractions, pelvic pain or cramping, abdominal pain or cramping, or any other concerns. Subjects will be counseled on avoidance of sexual intercourse and avoidance of overt exertion, yet, strict bed rest will not be advised. Subjects will be instructed to keep the "Patient Information Pamphlet" with them at all times while enrolled in this study. If patient either reports a lost or misplaced pamphlet at any point during the study or presents to any scheduled follow up appointment in the MFM clinic without the pamphlet, the patient will be provided with a new copy. The pamphlet includes a daily temperature log, an adverse/side effect log, and emergency contact information for key figures involved in this study. The pamphlet also includes a table in which dates and findings (i.e., EGA, maternal heart rate, fetal heart rate, maternal blood pressure, maternal temperature, and AFI) from follow-up MFM appointments are to be logged. The initial MFM follow-up appointment will be scheduled prior to discharge from the hospital for all subjects enrolled. Documentation of scheduled time and date will be noted on patient's discharge paperwork. Follow-up for both arms of the study will be scheduled within the MFM outpatient clinic weekly until subjects either reach 23 0/7 weeks gestation or show signs of change in clinical condition. Weekly follow-up visits will consist of vital signs (maternal heart rate, maternal blood pressure, temperature and weight), a physical examination of subject, an obstetric ultrasound to assess fetal well-being, calculate amniotic fluid index, and determine fetal heart rate, and weekly complete blood counts (lab draws). Patients will also be instructed to bring the antibiotic pill bottles the initial follow up appointment. The number of pills remaining will be counted to assess degree of antibiotic compliance. The results of these assessments, along with a copy of the "Patient Information Pamphlet", will be made at each follow up visit and stored within a data collection sheet. Each patient will be assigned an individual data collection sheet which will be marked with the patient's medical record number and unique subject identifier (determined as mentioned above).

All of the data collection sheets will be stored within a secure research binder. This binder will be kept secure in a locked desk drawer, within a locked office (MFM office located at 100 Woman's Way, Baton Rouge, LA 70817), when not in use. Access to study data will only be granted to Robert Clifton Moore, MD, Felicia LeMoine, MD, and Kaitlyn Taylor, MD during the study period. Following completion of the study, a final Excel spreadsheet will be created which will include all data previously collected, including the patient's unique identifier but excluding the patient's medical record number (de-identified). The final, compiled spreadsheet with de-identified data will be made available to Andrew Chapple, PhD for final data analysis. Upon completion of finalized data spreadsheet, the hard copies contained within the designated research binder will be disposed of in a secured, locked shred bin on Woman's Hospital campus. The spreadsheet will be encrypted and stored on an password-protected and encrypted laptop, property of the investigator Felicia LeMoine, MD. The spreadsheet will not be stored or saved onto any of the various, available internet storage services (i.e., DropBox, Google Drive, etc.)

If at any point during the study, subjects of either arm show signs of infection (fever, rigors, chills, pain), labor, abruption (vaginal bleeding), or fetal distress, subjects will be admitted to Woman's Hospital for induction of labor/delivery as recommended per established standards of care. Delivering physician will be either the patient's primary obstetrician or MFM specialist if subject received prenatal care at facility outside of Woman's Hospital.

If subject and the fetus show signs of continued stability with no adverse events/side effects, signs of chorioamnionitis, infection, labor, or placental abruption, from the time of rupture until 23 0/7 weeks gestation, the subject will be readmitted to Woman's Hospital's Labor and Delivery Unit at 23 0/7 for continued inpatient management until delivery. At the time of readmission, both treatment and control arms will receive fetal neuroprotective magnesium sulfate (6 gram loading dose, 6g in 100mL in-fused over 15- 20 minutes, followed by maintenance dose of 2g/hour at rate of 50mls/hr of 20g/500mL for a minimum of 12 hours), betamethasone course for fetal lung maturity (12mg intramuscular admin-istered every 24 hours for total of two doses), and latency antibiotics (a single dose of azithromycin 1g orally with 48-hour course of ampicillin 2g intravenously every 6 hours followed by amoxicillin 500mg orally every 9 hours for 5 days) as guided by current standard of care practices. Duration of treatment with magnesium sulfate will be standardized to a total of 12 hours on readmission and a plan for restart of medication if delivery is felt to imminent and at a gestational age of less than 34 weeks. While subjects are receiving magnesium sulfate, routine evaluations to assess for signs of magnesium toxicity will be performed as is outlined in the hospital policy regarding magnesium administration in pregnancy. Briefly this includes monitoring for signs and symptoms of magnesium overdose and therapy with calcium gluconate as need for magnesium toxicity.

Other orders to be instituted at the time of readmission include a repeat culture of urine, complete blood cell count, Maternal Fetal Medicine consultation, fetal ultrasound, regular diet, IV with saline lock, bed rest with bathroom privileges and fetal non-stress testing twice per day. Obstetric ultra-sounds will be repeated by the Maternal-Fetal medicine specialists within 24 hours of readmission and at least once every 7 days till delivery is indicated.

A rescue course of betamethasone (single dose of 12mg intramuscularly) will be administered if the subject does not deliver within 14 days of completion of the initial 2-dose course of betamethasone and if delivery is suspected within the next seven days.

Delivery following readmission will be at the discretion of the attending obstetrician in regards to evidence of maternal or fetal infection, labor, non-reassuring fetal assessment or placental abruption in addition to any other standard indication for delivery (ie., pre-eclampsia) or if patient reaches 34 0/7 weeks gestational age. Route of delivery will be determined by routine obstetrical indications.

All investigational products (study drugs) will be stored under appropriate storage conditions in a secure area according to local regulations. The investigator is responsible for ensuring that it is dispensed only to study subjects and only from official study sites by authorized personnel, as dictated by local regulations. The investigator is responsible for ensuring that the investigational product is stored under the appropriate environmental conditions (temperature, light, and humidity), as noted in the product labeling. Labels will be prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines for labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation
2. Gestational age of greater than 18 0/7 but less than or equal to 22 6/7
3. Diagnosis of prelabor premature rupture of membranes as determined by clinical examination noting either/or 1) visualization of amniotic fluid passing from the cervical canal and pooling in the vagina via sterile speculum examination, 2) a basic pH (i.e., positive nitrazine) test of vaginal fluid, 3) arborization (ferning) of dried vaginal fluid identified via microscopic examination, or 4) an amniotic fluid index (AFI) of less than 4cm
4. Greater than or equal to 18 years of age
5. Those with no known drug allergies or significant adverse reactions to azithromycin or amoxicillin
6. Afebrile at the time of presentation and throughout 24-hour observation period
7. Patient must be able to provide informed consent

Exclusion Criteria:

1. Fetal anomalies in current pregnancy
2. Diabetes mellitus, including both pre-gestational and gestational
3. Abnormal placentation
4. Poor dating with dating ultrasound performed later than or equal to 20 0/7 weeks
5. Current subchorionic hemorrhage or current vaginal bleeding on presentation
6. Hypertensive disease, including pre-gestational chronic hypertension, gestational hypertension and pre-eclampsia/eclampsia
7. History of amniocentesis during this pregnancy
8. History of cervical incompetence, history of cerclage in previous pregnancy or current cerclage in place
9. Current documented urinary tract infection or bacteriuria
10. Current documented genital tract infection (Chlamydia, gonorrhea, or trichomonas)
11. Immunocompromised (i.e., HIV positive, daily steroid use, or a history of autoimmune disease for which the patient is currently undergoing treatment with immunotherapy medication)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Latency period | Patient will be monitored from the date of diagnosis of previable prelabor rupture of membranes until date of delivery. This could vary from a duration of less than 1 day to 112 days.
  The number of days from diagnosis of previable prelabor rupture of membranes to the date of delivery

SECONDARY OUTCOMES:
Viability | Number of days from the time of rupture of membranes (earliest 18 0/7 weeks) to viability (23 0/7 weeks), max 35 days.
  The number of subjects in each arm that are able to reach 23 0/7 weeks gestational age following previable prelabor rupture of membranes between 18 0/7 and 22 6/7 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Moore, MD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will become available beginning 6 months after study publication and will be available indefinitely.
Access Criteria: Requests for data are available to all researchers; however, approval for access to data will be granted by primary investigator.

REFERENCES:
- [Background] Kilbride HW, Thibeault DW. Neonatal complications of preterm premature rupture of membranes. Pathophysiology and management. Clin Perinatol. 2001 Dec;28(4):761-85. doi: 10.1016/s0095-5108(03)00076-9. PMID 11817188
- [Background] Yeast JD. Preterm premature rupture of the membranes before viability. Clin Perinatol. 2001 Dec;28(4):849-60. doi: 10.1016/s0095-5108(03)00082-4. PMID 11758532
- [Background] Cunningham, F. G., MD, Leveno, K. J., MD, Dashe, J. S., MD, Hoffman, B. L., MD, Bloom, S. L., MD, Casey, B. M., MD, Spong, C. Y., MD (Eds.). (2014). Preterm Labor. In Williams Obstetrics(24th ed., pp. 848-849). New York, NY: McGraw Hill Education.
- [Background] Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Ramsey RD, Rabello YA, Meis PJ, Moawad AH, Iams JD, Van Dorsten JP, Paul RH, Bottoms SF, Merenstein G, Thom EA, Roberts JM, McNellis D. Antibiotic therapy for reduction of infant morbidity after preterm premature rupture of the membranes. A randomized controlled trial. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. JAMA. 1997 Sep 24;278(12):989-95. PMID 9307346
- [Background] Mercer BM, Goldenberg RL, Das AF, Thurnau GR, Bendon RW, Miodovnik M, Ramsey RD, Rabello YA; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. What we have learned regarding antibiotic therapy for the reduction of infant morbidity after preterm premature rupture of the membranes. Semin Perinatol. 2003 Jun;27(3):217-30. doi: 10.1016/s0146-0005(03)00016-8. PMID 12889589
- [Background] American College of Obstetricians and Gynecologists; Society for Maternal-Fetal Medicine. Obstetric Care consensus No. 6: Periviable Birth. Obstet Gynecol. 2017 Oct;130(4):e187-e199. doi: 10.1097/AOG.0000000000002352. PMID 28937572
- [Background] Antenatal corticosteroids revisited: repeat courses. NIH Consens Statement. 2000 Aug 17-18;17(2):1-18. PMID 11725806
- [Background] Doyle LW, Crowther CA, Middleton P, Marret S, Rouse D. Magnesium sulphate for women at risk of preterm birth for neuroprotection of the fetus. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD004661. doi: 10.1002/14651858.CD004661.pub3. PMID 19160238
- [Background] Mercer BM, Crocker LG, Boe NM, Sibai BM. Induction versus expectant management in premature rupture of the membranes with mature amniotic fluid at 32 to 36 weeks: a randomized trial. Am J Obstet Gynecol. 1993 Oct;169(4):775-82. doi: 10.1016/0002-9378(93)90004-3. PMID 8238131
- [Background] Broekhuizen FF, Gilman M, Hamilton PR. Amniocentesis for gram stain and culture in preterm premature rupture of the membranes. Obstet Gynecol. 1985 Sep;66(3):316-21. PMID 2410839
- [Background] Cotton DB, Hill LM, Strassner HT, Platt LD, Ledger WJ. Use of amniocentesis in preterm gestation with ruptured membranes. Obstet Gynecol. 1984 Jan;63(1):38-43. PMID 6691016
- [Background] Zlatnik FJ, Cruikshank DP, Petzold CR, Galask RP. Amniocentesis in the identification of inapparent infection in preterm patients with premature rupture of the membranes. J Reprod Med. 1984 Sep;29(9):656-60. PMID 6492031
- [Background] Mercer BM, Moretti ML, Prevost RR, Sibai BM. Erythromycin therapy in preterm premature rupture of the membranes: a prospective, randomized trial of 220 patients. Am J Obstet Gynecol. 1992 Mar;166(3):794-802. doi: 10.1016/0002-9378(92)91336-9. PMID 1550145
- [Background] Romero R, Emamian M, Quintero R, Wan M, Hobbins JC, Mazor M, Edberg S. The value and limitations of the Gram stain examination in the diagnosis of intraamniotic infection. Am J Obstet Gynecol. 1988 Jul;159(1):114-9. doi: 10.1016/0002-9378(88)90503-0. PMID 2456013
- [Background] Oh KJ, Lee KA, Sohn YK, Park CW, Hong JS, Romero R, Yoon BH. Intraamniotic infection with genital mycoplasmas exhibits a more intense inflammatory response than intraamniotic infection with other microorganisms in patients with preterm premature rupture of membranes. Am J Obstet Gynecol. 2010 Sep;203(3):211.e1-8. doi: 10.1016/j.ajog.2010.03.035. Epub 2010 Aug 3. PMID 20678747
- [Background] DiGiulio DB, Romero R, Kusanovic JP, Gomez R, Kim CJ, Seok KS, Gotsch F, Mazaki-Tovi S, Vaisbuch E, Sanders K, Bik EM, Chaiworapongsa T, Oyarzun E, Relman DA. Prevalence and diversity of microbes in the amniotic fluid, the fetal inflammatory response, and pregnancy outcome in women with preterm pre-labor rupture of membranes. Am J Reprod Immunol. 2010 Jul 1;64(1):38-57. doi: 10.1111/j.1600-0897.2010.00830.x. Epub 2010 Mar 21. PMID 20331587
- [Background] Svigos, John M, et al. "Chapter 63: Prelabor Rupture of Membranes." High Risk Pregnancy: Management Options - Expert Consult, by David K. James et al., Saunders, 2010, pp. 1321-132.
- [Background] Amsden GW. Erythromycin, clarithromycin, and azithromycin: are the differences real? Clin Ther. 1996 Jan-Feb;18(1):56-72; discussion 55. doi: 10.1016/s0149-2918(96)80179-2. PMID 8851453
- [Background] Heikkinen T, Laine K, Neuvonen PJ, Ekblad U. The transplacental transfer of the macrolide antibiotics erythromycin, roxithromycin and azithromycin. BJOG. 2000 Jun;107(6):770-5. doi: 10.1111/j.1471-0528.2000.tb13339.x. PMID 10847234
- [Background] Esteves JS, de Sa RA, de Carvalho PR, Coca Velarde LG. Neonatal outcome in women with preterm premature rupture of membranes (PPROM) between 18 and 26 weeks. J Matern Fetal Neonatal Med. 2016;29(7):1108-12. doi: 10.3109/14767058.2015.1035643. Epub 2015 Jul 3. PMID 26138545
- [Background] Manuck TA, Eller AG, Esplin MS, Stoddard GJ, Varner MW, Silver RM. Outcomes of expectantly managed preterm premature rupture of membranes occurring before 24 weeks of gestation. Obstet Gynecol. 2009 Jul;114(1):29-37. doi: 10.1097/AOG.0b013e3181ab6fd3. PMID 19546755
- [Background] Schucker JL, Mercer BM. Midtrimester premature rupture of the membranes. Semin Perinatol. 1996 Oct;20(5):389-400. doi: 10.1016/s0146-0005(96)80006-1. PMID 8912993
- [Background] Linehan LA, Walsh J, Morris A, Kenny L, O'Donoghue K, Dempsey E, Russell N. Neonatal and maternal outcomes following midtrimester preterm premature rupture of the membranes: a retrospective cohort study. BMC Pregnancy Childbirth. 2016 Jan 29;16:25. doi: 10.1186/s12884-016-0813-3. PMID 26831896
- [Background] Deutsch A, Deutsch E, Totten C, Downes K, Haubner L, Belogolovkin V. Maternal and neonatal outcomes based on the gestational age of midtrimester preterm premature rupture of membranes. J Matern Fetal Neonatal Med. 2010 Dec;23(12):1429-34. doi: 10.3109/14767051003678069. Epub 2010 Mar 17. PMID 20233131
- [Background] Moore T, Hennessy EM, Myles J, Johnson SJ, Draper ES, Costeloe KL, Marlow N. Neurological and developmental outcome in extremely preterm children born in England in 1995 and 2006: the EPICure studies. BMJ. 2012 Dec 4;345:e7961. doi: 10.1136/bmj.e7961. PMID 23212880
- See also: Werth, Brian. "Macrolides - Infectious Diseases." Merck Manuals Professional Edition, July 2018 — https://www.merckmanuals.com/professional/infectious-diseases/bacteria-and-antibacterial-drugs/macrolides#v1604552.
- See also: LabCorp. (2018). Wet Prep. Retrieved December 30, 2018 — https://www.labcorp.com/test-menu/36906/wet-prep
- See also: LabCorp. (2018). Complete Blood Count (CBC) with Differential. Retrieved December 30, 201 — https://www.labcorp.com/test-menu/23041/complete-blood-count-cbc-with-differentia
- See also: LabCorp. (2018). Group B Streptococcus Colonization Detection Culture. Retrieved December 30, 2018 — https://www.labcorp.com/test-menu/26276/group-b-istreptococcus-i-colonization-detection-culture

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04047849/Prot_000.pdf
  • Informed Consent Form (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04047849/ICF_001.pdf